CLINICAL TRIAL: NCT00684541
Title: Interpretation Modification Program for Social Phobia
Acronym: SP Interp
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: San Diego State University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Nader Amir, Professor, San Diego State University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1-Amir; 5R34MH073004-03 (NIH)
Record Dates: First submitted 2008-05-22; First posted 2008-05-26 (Estimated); Results first posted 2014-05-01 (Estimated); Last update posted 2014-05-01 (Estimated); Status verified 2014-04

CONDITIONS: Social Anxiety Disorder; Social Phobia
Keywords: Social Anxiety; Information Processing; Interpretation
MeSH Terms: conditions — Phobia, Social

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Interpretation Modification Program (Experimental): The IMP procedure was identical to the word-sentence association paradigm (WSAP; Beard & Amir, 2009) except participants received feedback about their responses. Participants received positive feedback when they endorsed benign interpretations or rejected threat interpretations of the ambiguous sentences on 100% of trials and negative feedback when they endorsed threat interpretations or rejected benign interpretations on 100% of trials. This feedback manipulation was intended to reinforce a benign interpretation bias and extinguish the threat interpretation bias. Participants completed two blocks of 110 training trials in each session. Participants who completed Set A during the WSAP assessment saw Set B during the IMP and vice versa. Each IMP session lasted approximately 20 min.
  Interventions: Behavioral: Interpretation Modification Program
- Interpretation Control Condition (Placebo Comparator): The ICC was identical to the IMP, except that participants received positive feedback when they endorsed threat interpretations on half (50%) of the trials and negative feedback when they endorsed threat interpretations for the remaining half (50%) of trials. This frequency was the same for benign interpretations. Thus, the control group was reinforced equally for making threat and benign interpretations. The ICC was not intended to change interpretation significantly in either direction.
  Interventions: Behavioral: Interpretation Control Condition

INTERVENTIONS:
Behavioral: Interpretation Modification Program — The IMP protocol includes twelve 30-min sessions delivered over a 6-week period. Each session will comprise 220 trials. In each trial, participants will first see either a non-threat or a threat (e.g. "graceful" or "clumsy") word on the computer screen. They will then see an ambiguous sentence (e.g. "You dance at the party") and will be asked to indicate if the word and sentence were related by pressing a corresponding key. Participants will receive positive feedback (i.e., "You are correct!") when they endorse a non-threat interpretation or reject a threat interpretation of an ambiguous sentence. Participants will receive negative feedback (i.e., "You are incorrect.") when they endorse a threat interpretation or reject a non-threat interpretation of an ambiguous sentence.
  Arms: Interpretation Modification Program
Behavioral: Interpretation Control Condition — Participants assigned to the PC completed an identical procedure to the IMP procedure except that feedback about participants' performance was not contingent on the type of interpretation (i.e., non-threat or threat) endorsed. Thus, participants in the PC received positive feedback 50% of the time when viewing a threat interpretation and 50% of the time when viewing a non-threat interpretation.
  Arms: Interpretation Control Condition

SUMMARY:
Generalized Social Phobia is characterized by severe social anxiety that leads to functional impairment (Schneider et al., 1992). Despite its high prevalence, many individuals do not receive treatment or are unresponsive to current therapies. Thus there is a clear need to continue to develop highly effective and efficient treatments for social phobia. This three year project aims to test a computerized treatment for social phobia in a double-blind, placebo-controlled study designed to modify interpretation biases that may maintain anxiety.

DETAILED DESCRIPTION:
Social phobia is characterized by severe social anxiety leading to functional impairment (Schneider et al., 1992). Despite its high prevalence (13%, Kessler et al., 1994) over 30% of individuals with social anxiety who need treatment do not receive treatment (Olfson, et al., 2000) and 40% of individuals who present for treatment do not respond (39%, Heimberg, et al., 1998; 42%, Liebowitz et al., 2005). Thus, there is a clear need to develop highly effective and efficient treatments for GSP. Reducing negative interpretation of social events is an efficacious treatment for SP because:

1. benign interpretations is associated with improvement in social anxiety after treatment (e.g., Franklin, Huppert, Langner, Leiberg, & Foa, 2005)
2. negative interpretations are implicated in the pathogenesis of SP (e.g., Rapee & Heimberg, 1997)
3. SPs have more negative interpretations of social events than non-anxious controls and individuals with other anxiety disorders (e.g., Amir et al, 1998)
4. this bias ameliorates after successful treatment (e.g., Stopa & Clark, 2000).

Therefore, changing negative interpretations is an efficacious treatment for SP, and current cognitive-behavioral therapies use cognitive restructuring (CR) to target negative interpretations and replace them with more benign interpretations (Heimberg, et al., 1998). The goal of the current proposal is to test a new computerized treatment for SP that is designed to change negative interpretations. We chose a computerized intervention to increase efficiency and ease of delivery. We chose to test this intervention in GSP because interpretation bias is especially relevant to this clinical population. The long-term goal of this project is to improve service delivery using a widely available and economical intervention for GSP. More specifically, we will test three hypotheses in this proposal:

1. Individuals with GSP completing the Interpretation Modification Program (IMP) will show a reduction in their negative interpretation
2. Participants in the IMP will show a decrease in their social anxiety symptoms
3. Change in social anxiety symptoms will be mediated by the change in interpretation scores, suggesting that interpretation change reduced social anxiety symptoms.

Pilot data (n=34) suggest that this intervention is efficacious. Thus, we aim to develop further and validate this highly efficient treatment for changing interpretations as a cost-effective treatment for patients with social phobia.

ELIGIBILITY:
Inclusion Criteria:

* Principle DSM-IV-TR (APA, 2000) Diagnosis of social phobia - Generalized Type (GSP)

Exclusion Criteria:

* No change in medication type or dosage twelve weeks prior to initiating treatment
* No current psychotherapy
* No evidence of suicidal intent
* No evidence of substance abuse in the last 6 months
* No evidence of current or past schizophrenia, bipolar disorder, or organic mental disorder

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2007-09; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nader Amir, Ph.D., Principal Investigator — SDSU/UCSD
Locations (1):
- San Diego State University, San Diego, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Interpretation Modification Program (IMP): The IMP procedure was identical to the word-sentence association paradigm (WSAP; Beard & Amir, 2009) except that participants received feedback about their responses. Specifically, participants received positive feedback when they endorsed benign interpretations or rejected threat interpretations of the ambiguous sentences on 100% of trials. Participants received negative feedback when they endorsed threat interpretations or rejected benign interpretations on 100% of trials. This feedback manipulation was intended to reinforce a benign interpretation bias and extinguish the threat interpretation bias. Participants completed two blocks of 110 training trials (76 social and 34 nonsocial) in each session. Participants who completed Set A during the WSAP assessment saw Set B during the IMP and vice versa. Thus, participants were assessed with different materials than those seen during the IMP. Each IMP session lasted approximately 20 min.
- Interpretation Control Condition (ICC): The ICC was identical to the IMP, except that participants received positive feedback when they endorsed threat interpretations on half (50%) of the trials and negative feedback when they endorsed threat interpretations for the remaining half (50%) of trials. This frequency was the same for benign interpretations. Thus, the control group was reinforced equally for making threat and benign interpretations. The ICC was not intended to change interpretation significantly in either direction.
Period: Overall Study
Arm/Group | Interpretation Modification Program (IMP) | Interpretation Control Condition (ICC)
Started | 23 | 26
Completed | 20 | 23
Not Completed | 3 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Interpretation Modification Program | Interpretation Control Condition | Total
Number analyzed (Participants) | 23 | 26 | 49
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 23 | 26 | 49
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 16 | 35
  Male | 4 | 10 | 14
Region of Enrollment [Number; unit: participants]
  United States | 23 | 26 | 49

OUTCOME MEASURES:

1. Primary Outcome: Liebowitz Social Anxiety Scale (LSAS)
Description: Our primary outcome measure was the clinician-administered LSAS (Liebowitz, 1987), a 24-item scale that provides separate scores for fear and avoidance of social interaction and performance situations. LSAS scores range from 0 to 144. The LSAS has strong psychometric properties (Heimberg et al., 1999) and is arguably the gold-standard outcome measure in treatment research in SAD (e.g., Clark et al., 2006; Heimberg et al., 1998). Higher scores indicate more severe symptoms.
Time Frame: Pre, Post (6 weeks), Followup (3 months after post-assessment)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Interpretation Modification Program | Interpretation Control Condition
Number analyzed (Participants) | 20 | 23
units on a scale
  pre-tx | 82.0 (18.4) | 77.7 (18.6)
  post | 50.2 (19.3) | 67.6 (26.2)
  follow-up | 40.8 (21.6) | NA (NA) — Data not collected for ICC at follow-up.

2. Secondary Outcome: Social Phobia and Agoraphobia Inventory
Description: Our secondary outcome assessment of social anxiety symptoms was the Social Phobia and Anxiety Inventory (SPAI; Turner, Beidel, Dancu, & Stanley, 1989), a 45-item self-rated measure that assesses the cognitive, behavioral, and somatic dimensions of SAD. SPAI scores range from 45 to 315, with higher scores indicating more severe symptoms. Previous research suggests that the SPAI has sound psychometric properties (e.g., Turner et al., 1989). Internal consistencies for these measures in the current sample were satisfactory.
Time Frame: Pre, Post (6 weeks), Followup (3 months after post-assessment)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Interpretation Modification Program | Interpretation Control Condition
Number analyzed (Participants) | 23 | 26
units on a scale
  pre-tx | 145.0 (26.8) | 146.1 (21.8)
  post-tx | 112.0 (34.4) | 118.1 (43.7)
  follow-up | 94.7 (37.7) | NA (NA) — Data not collected from ICC group at follow-up

ADVERSE EVENTS:
Arm/Group | Interpretation Modification Program | Interpretation Control Condition
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/26
Other Adverse Events (participants affected / at risk) | 0/23 | 0/26

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No